CLINICAL TRIAL: NCT00243529
Title: In Vivo Responses of DC Vaccines Presenting HLA Class I and II Restricted Tumor Epitopes Either by Peptide-pulsing or mRNA Transfection in Melanoma Patients
Brief Title: Peptide-pulsed vs. RNA-transfected Dendritic Cell Vaccines in Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Prof. C.J.A. Punt, MD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-2917; KWF 2003-2917
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-02

CONDITIONS: Melanoma Stage III or IV
Keywords: Dendritic cells; Melanoma; Vaccine; Immunotherapy; RNA; Peptides
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MHC Class I restricted epitopes (Active Comparator): HLA-A2.1 patients are vaccinated with dendritic cells loaded with MHC Class I restricted epitopes of tumor antigens gp100 and tyrosinase
  Interventions: Biological: autologous dendritic cell vaccine
- MHC Class I and II restricted epitopes (Experimental): HLA-A2.1 and HLA-DR4 patients are vaccinated with dendritic cells loaded with MHC Class I and II restricted epitopes of tumor antigens gp100 and tyrosinase
  Interventions: Biological: autologous dendritic cell vaccine
- mRNA transfected DC (Experimental): HLA-A2.1 and/or HLA-DR4 patients are vaccinated with dendritic cells transfected with mRNA encoding tumor antigens gp100 and tyrosinase
  Interventions: Biological: autologous dendritic cell vaccine

INTERVENTIONS:
Biological: autologous dendritic cell vaccine

SUMMARY:
Dendritic cells (DCs)are the most potent antigen-presenting cells of the immune system, as such they are able to direct the immune system specifically against cancer cells. Currently DCs are used in clinical vaccination studies and immunological and clinical responses have been observed. For inducing anti-tumor immunity, the DCs have to be loaded with tumor antigen (i.e. molecular structures that are presented by the tumor, that are recognized by the immune system). Currently most studies use tumor peptides (small protein fragments) for this purpose. This approach has several disadvantages: only patients with a certain HLA-type can be treated and the immune response that is induced by the vaccine is limited to the used peptides. These disadvantages do not exist when the DCs present antigen which is endogenously processed, for example after RNA transfection. For this reason we investigate the immunogenicity of DCs that are pulsed with peptides or transfected with mRNA encoding melanoma associated antigens in stage III and IV melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

For both stage III and IV

* Histological proof of cutaneous melanoma
* Melanoma expressing both gp100 and tyrosinase, each in approximately 20% or more of cells by immunohistochemistry staining,
* HLA type A2 and/or A3, with known HLA-DR4 expression,
* WBC > 3.0 x 109/l, lymphocytes > 0.8 x 109/l, platelets > 100 x 109/l, serum creatinine < 150 μmol/l, serum bilirubin < 25 μmol/l.
* Expected adequacy of follow-up,
* Written informed consent.

For Stage III only

* Stage III melanoma according to the 2001 AJCC criteria.
* Start of treatment within 2 months of lymph node dissection for melanoma stage III

For stage IV only

-Stage IV melanoma according to the 2001 AJCC criteria. Limited tumor burden; LDH < 2x upper limit of normal

Exclusion Criteria:

For both stage III and IV

* No autoimmune disorders, no concomitant use of immunosuppressive drugs,
* no serious concomitant disease, no serious active infections, no other malignancy in the past 5 years with the exception of curatively treated carcinoma in-situ of the cervix/squamous cell carcinoma of the skin,
* No known allergy to shell fish (contains KLH) are excluded.
* No pregnancy or lactation,

For stage III only:

* No signs or symptoms of distant metastases as defined by normal history, physical examination, chest X-ray and serum LDH.
* No concomitant or previous systemic treatment for melanoma

For stage IV only:

* No clinical signs of CNS metastases, in patients with a clinical suspicion of CNS metastases, a CT scan of the brain should be performed to exclude this.
* No prior chemotherapy, immunotherapy, or radiotherapy within three months before planned vaccination is allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-04; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Immune response | first 10 years

SECONDARY OUTCOMES:
Safety | first 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Prof. C.J.A. Punt, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Center; Prof. G.J. Adema, PhD, Principal Investigator — Radboud University Nijmegen Medical Center/Nijmegen Center for Molecular Life Sciences
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, PO Box 9101, Netherlands

REFERENCES:
- [Background] de Vries IJ, Bernsen MR, Lesterhuis WJ, Scharenborg NM, Strijk SP, Gerritsen MJ, Ruiter DJ, Figdor CG, Punt CJ, Adema GJ. Immunomonitoring tumor-specific T cells in delayed-type hypersensitivity skin biopsies after dendritic cell vaccination correlates with clinical outcome. J Clin Oncol. 2005 Aug 20;23(24):5779-87. doi: 10.1200/JCO.2005.06.478. PMID 16110035
- [Background] Lesterhuis WJ, de Vries IJ, Adema GJ, Punt CJ. Dendritic cell-based vaccines in cancer immunotherapy: an update on clinical and immunological results. Ann Oncol. 2004;15 Suppl 4:iv145-51. doi: 10.1093/annonc/mdh919. No abstract available. PMID 15477299
- [Background] Figdor CG, de Vries IJ, Lesterhuis WJ, Melief CJ. Dendritic cell immunotherapy: mapping the way. Nat Med. 2004 May;10(5):475-80. doi: 10.1038/nm1039. PMID 15122249
- [Background] de Vries IJ, Lesterhuis WJ, Scharenborg NM, Engelen LP, Ruiter DJ, Gerritsen MJ, Croockewit S, Britten CM, Torensma R, Adema GJ, Figdor CG, Punt CJ. Maturation of dendritic cells is a prerequisite for inducing immune responses in advanced melanoma patients. Clin Cancer Res. 2003 Nov 1;9(14):5091-100. PMID 14613986
- [Background] De Vries IJ, Krooshoop DJ, Scharenborg NM, Lesterhuis WJ, Diepstra JH, Van Muijen GN, Strijk SP, Ruers TJ, Boerman OC, Oyen WJ, Adema GJ, Punt CJ, Figdor CG. Effective migration of antigen-pulsed dendritic cells to lymph nodes in melanoma patients is determined by their maturation state. Cancer Res. 2003 Jan 1;63(1):12-7. PMID 12517769
- [Background] de Vries IJ, Eggert AA, Scharenborg NM, Vissers JL, Lesterhuis WJ, Boerman OC, Punt CJ, Adema GJ, Figdor CG. Phenotypical and functional characterization of clinical grade dendritic cells. J Immunother. 2002 Sep-Oct;25(5):429-38. doi: 10.1097/00002371-200209000-00007. PMID 12218781
- [Background] Adema GJ, de Vries IJ, Punt CJ, Figdor CG. Migration of dendritic cell based cancer vaccines: in vivo veritas? Curr Opin Immunol. 2005 Apr;17(2):170-4. doi: 10.1016/j.coi.2005.01.004. PMID 15766677
- See also: Home page of the Radboud University Nijmegen Medical Centre — http://www.umcn.nl